CLINICAL TRIAL: NCT02351765
Title: A Phase Ib, Multi-centre, Open-label Study of a First-in-class Nucleotide Analogue Acelarin (NUC-1031) in Combination With Cisplatin in Patients With Locally Advanced/Metastatic Biliary Tract Cancers
Brief Title: ABC-08: Phase Ib Trial of Acelarin in Combination With Cisplatin in Locally Advanced/ Metastatic Biliary Tract Cancers
Acronym: ABC-08
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFTSp096; 2015-000100-26 (EudraCT Number)
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Biliary Tract Cancer; Gallbladder Cancer; Cholangiocarcinoma; Ampullary Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms; Gallbladder Neoplasms; Cholangiocarcinoma | interventions — NUC-1031; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Acelarin & Cisplatin (Experimental): The maximum tolerated dose (MTD) of Acelarin in combination with 25mg/m2 Cisplatin will be determined.
  The starting dose will be 625mg/m2 Acelarin which will be escalated to 725mg/m2 if the criteria for dose escalation is met (i.e. the proportion of dose limiting toxicities is acceptable as detailed in the protocol). Escalation will continue in accordance with the protocol up to a maximum of 925mg/m2. Only if the MTD is exceeded at the starting dose level (at least 2 of 3 participants or at least 2 of 6 participants have DLT at the first dose level) will there be a de-escalation to 500mg.
  Interventions: Drug: Acelarin; Drug: Cisplatin

INTERVENTIONS:
Drug: Acelarin — First-in-class nucleotide analogue
  Other Names: Code name: NUC-1031
Drug: Cisplatin — Platinum-compound chemotherapy drug
  Other Names: Anatomical Therapeutic Chemical (ATC) code: L01XA01

SUMMARY:
The purpose of this study is to determine the recommended phase II dose, and to assess the safety of acelarin in combination with cisplatin in patients with locally advanced/ metastatic biliary tract cancers.

DETAILED DESCRIPTION:
Active chemotherapy drugs for the treatment of advanced biliary tract cancers (ABC) include gemcitabine, fluoropyrimidines and platinum agents. The United Kingdom (UK) National Cancer Research Network (NCRN) ABC-02 study established cisplatin and gemcitabine as the standard of care for the first-line treatment of patients with ABC and this regimen has been widely adopted in the UK and internationally. However, inherent and acquired tumour resistance limits the efficacy of gemcitabine and it is necessary to explore alternative treatments.

The study will explore the combination of acelarin, a drug designed to specifically overcome the key cancer resistance mechanisms associated with gemcitabine, with cisplatin. As this is the first time the combination of acelarin and cisplatin will be given to patients the aim of the study is to investigate the safety of the combination and to establish the recommended phase II dose of acelarin.

This is a phase Ib, single-arm, multi-centre, open-label trial. The trial design is a classic 3+3 design where patients are recruited into cohorts of 3 to 6 patients at different dose levels until the dose level for phase II is determined. Patients in each cohort will be monitored closely for safety and drug toxicity.

Secondary trial objectives will involve assessing the activity of acelarin in combination with cisplatin in terms of; progression-free survival, overall survival and response rate, as well as exploring the pharmacokinetic profile of the combination.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically verified, non-resectable or recurrent/metastatic cholangiocarcinoma, gallbladder or ampullary carcinoma.
* No prior systemic therapy allowed for advanced biliary cancer. Prior low dose chemotherapy used with or without radiotherapy in the adjuvant setting is allowed if completed > 6 months from enrolment. Recent palliative radiation (within 28 days prior to consent) is allowed if candidate has measurable disease outside radiation field.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Age ≥ 18 years and life expectancy > 3 months.
* Adequate renal function with serum urea and serum creatinine < 1.5 times upper limit of normal (ULN) and creatinine clearance ≥ 30ml/min.
* Adequate haematological function: Hb ≥ 10g/dl, white blood count (WBC) ≥ 3.0 x 10*9/L, absolute neutrophil count (ANC) ≥ 1.5 x 10*9/L, platelet count ≥ 100,000/mm3.
* Adequate liver function: total bilirubin < 30 μmol/L and alkaline phosphatase, along with aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≤ 5 x ULN.
* Adequate biliary drainage, with no evidence of ongoing infection.
* Women of child bearing age MUST have a negative pregnancy test prior to study entry AND be using a highly effective contraception method (combined or progestogen-only hormonal contraception, intrauterine device, intrauterine hormone-releasing system, vasectomised partner*(a) or sexual abstinence**(b)) which must be continued for 6 months after the end of study treatment, unless child bearing potential has been terminated by surgery/radical radiotherapy or infertility due to bilateral tubal occlusion.
* Male subjects must either have had a successful vasectomy (confirmed azoospermia) or they and their female partner meet the criteria above (not of childbearing potential or practicing adequate contraception [e.g. combined or progestogen-only hormonal contraception, intrauterine device, intrauterine hormone-releasing system, sexual abstinence**(b)] throughout the study period and for 6 months after the end of study treatment).
* Patients must not have a history of other malignant diseases (within the previous 5 years and there must be no evidence of recurrence), other than adequately treated non-melanotic skin cancer or in-situ carcinoma of the uterine cervix.
* Patients must have given written informed consent.

  * (a) The vasectomised partner must have received medical assessment confirming surgical success.

    * (b) Sexual abstinence in line with the preferred and usual lifestyle of the subject.

Exclusion Criteria:

* History of allergic reactions attributed to previous gemcitabine or cisplatin treatment.
* Documented history of allergic reactions attributed to any of the excipients used in the formulation (Kolliphor ELP; Tween 80; DMA).
* Previous treatment with Acelarin.
* Incomplete recovery from previous therapy (surgery/adjuvant therapy/radiotherapy) or unresolved biliary tree obstruction.
* Any evidence of severe or uncontrolled systemic diseases which, in the view of the investigator, makes it undesirable for the patient to participate in the trial.
* Evidence of significant clinical disorder or laboratory finding which, in the opinion of the investigator makes it undesirable for the patient to participate in the trial.
* Any patient with a medical or psychiatric condition that impairs their ability to give informed consent.
* Any other serious uncontrolled medical conditions.
* Clinical evidence of metastatic disease to the brain.
* Any pregnant or lactating woman.
* Pre-existing hearing impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-01; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Safety profile of Acelarin in combination with Cisplatin, assessed by total incidence and rate of grade 3 and 4 adverse events according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) | Adverse events recorded from initiation of therapy until 30 day post-treatment
  Safety will be assessed by comparing the total incidence and rate of grade 3 and 4 adverse events that occur after initiation of therapy, according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)
Maximum Tolerated Dose (MTD) of Aclerain in combination with Cisplatin | After 13 months of first patient included
  The MTD will be defined as the maximum dose level at which 0/3 patients or 1/6 patients experience dose-limiting toxicity (DLT). At any dose level, DLT in 1/3 patients will lead to expansion to 6 patients. If 2/6 patients experience DLT the preceding dose level will be declared the MTD. At the MTD up to 6 additional patients may be enrolled. If this level is well tolerated, it will be declared the recommended phase II dose (RP2D).

SECONDARY OUTCOMES:
Progression-free survival | Evaluated by 6 weekly follow-up until 12 months after the last patient included
  Clinical progression assessed every six weeks, radiological progression assessed to Response Evaluation Criteria in Solid Tumors (RECIST) criteria every 12 weeks.
Overall survival | Evaluated by 6 weekly follow-up until 12 months after the last patient included
Response rate | After 12 weeks of treatment
  Response will be calculated as a composite of objective response rate (ORR) by RECIST 1.1 (summation of patients with a complete or partial response [any time]).
Exploration of the pharmacokinetic profile for the combination of Acelarin with Cisplatin | At baseline (prior to chemotherapy administration), 30, 60 and 240 minutes following line flush at the end of acelarin administration. Cycle 1 day 1 only
  Plasma and intracellular levels of acelarin, cisplatin, gemcitibine (2', 2'-difluoro 2'-deoxycytidine) (dFdC), gemcitabine monophosphate (dFdCMP), gemcitabine diphosphate (dFdCDP), gemcitabine triphosphate (dFdCTP) and difluorodeoxyuridine (dFdU) will be measured and correlated with clinical activity and safety profile.

CONTACTS AND LOCATIONS:
Overall Officials: Mairéad G McNamara, MD, Study Chair — The Christie NHS Foundation Trust
Locations (5):
- United Kingdom (5):
  - Beatson Oncology Centre, Glasgow
  - Clatterbridge Cancer Centre, Liverpool
  - Imperial College London, London
  - University College London, London
  - The Christie NHS Foundation Trust, Manchester

REFERENCES:
- [Derived] McNamara MG, Bridgewater J, Palmer DH, Faluyi O, Wasan H, Patel A, Ryder WD, Barber S, Gnanaranjan C, Ghazaly E, Evans TRJ, Valle JW. A Phase Ib Study of NUC-1031 in Combination with Cisplatin for the First-Line Treatment of Patients with Advanced Biliary Tract Cancer (ABC-08). Oncologist. 2021 Apr;26(4):e669-e678. doi: 10.1002/onco.13598. Epub 2020 Dec 3. PMID 33210382